CLINICAL TRIAL: NCT01408095
Title: A 12-Week, Phase 2, Randomized, Double-Blind, Active-Controlled Study of LY2608204 Given as Monotherapy or in Combination With Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study in Patients With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated no patients were screened or enrolled
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14090; I3P-MC-GKBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; glimepiride; diabetes type II; diabetes type 2; Type 2 diabetes; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — globalagliatin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2608204 (Experimental): 80 to 400 mg, Doses will be titrated to reach glycemic targets during the first 4 weeks. The starting dose level depends on the participant's HbA1c level measured at Screening. Administered orally, daily for 12 weeks
  Interventions: Drug: LY2608204
- Glimepiride (Active Comparator): 1 to 6 mg, Doses will be titrated to reach glycemic targets during the first 4 weeks. Administered orally, daily for 12 weeks
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: LY2608204 — Administered orally
  Arms: LY2608204
Drug: Glimepiride — Administered orally
  Arms: Glimepiride

SUMMARY:
The study is designed to see if once daily oral dosing of LY2608204 will help control diabetes as measured by the glycosylated fraction of hemoglobin A (HbA1c) level. It will also help to determine the safety of the medication and the most useful doses of the medication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus prior to entering the trial
* May be treated with:

  1. Diet and exercise alone or
  2. Diet and exercise in combination with a stable dose of metformin for at least 3 months before Screening or
  3. Diet and exercise in combination with a stable dose of sulfonylurea or meglitinide (repaglinide, nateglinide) for at least 3 months before Screening or
  4. Diet and exercise in combination with stable doses of metformin and sulfonylurea or metformin and meglitinides for at least 3 months before Screening and have had diabetes for at least 6 years
* Must have an Hemoglobin A1c value between 7% and 10%
* Must have a body mass index (BMI) between 20 and 40 kg/m2
* Must have stable weight during the 3 months prior to Screening (weight change not to exceed 5 kg (11 lb))
* If female, you must not be able to get pregnant
* Must be well motivated, capable, and willing to complete study required glucose monitoring and instruction

Exclusion Criteria:

* Use of insulin or any antidiabetic agent other than metformin or sulfonylurea or meglitinide during the 3 months prior to Screening
* Have a gastrointestinal disease that significantly impacts gastric emptying or motility or have undergone gastric bypass or gastric banding surgery
* Have had more than one episode of severe hypoglycemia within 6 months prior to entry into the study, or are currently diagnosed as having hypoglycemia unawareness or have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months
* Are currently taking or have taken within the last 2 months, prescription or over-the counter medications which affect body weight
* Have cardiac disease with functional status that is New York Heart Association [NYHA] Class II, III, or IV or a history of myocardial infarction, unstable angina, or decompensated congestive heart failure in the past 6 months.
* Have poorly controlled hypertension, history of malignant hypertension, evidence of renal artery stenosis and/or evidence of labile blood pressure including symptomatic postural hypotension. Doses of antihypertensive medications must be stable for 30 days before randomization
* Have a QTcB (Bazett's-corrected QT interval) interval greater than 450 msec for men or greater than 470 for women at Screening or any personal history of ventricular tachycardia or unexplained syncope
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or significantly elevated liver blood tests
* Are currently receiving renal dialysis, have a serum creatinine greater than 2.0 mg/dL (177 μmol/L) or a calculated creatinine clearance of less than 60 ml/min or in patients being treated with metformin, have other known contradictions to metformin use including, but not limited to, a serum creatinine above (or creatinine clearance below) what is approved in the metformin product label
* Have fasting state hypertriglyceridemia (defined as greater than 5.65 mmol/L, 500 mg/dl) at Screening. If taking lipid-lowering agents, doses of these medications must be stable for 30 days prior to randomization.
* Are receiving chronic (for more than 2 weeks) systemic glucocorticoid therapy (excluding topical or inhaled preparations) or have received such therapy within 4 weeks immediately prior to Randomization
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* Have a history of seizure disorder
* Are currently using or intend to use inhibitors of Cytochrome P450 family 3A (CYP3A4)
* Currently taking a medication that is a sensitive substrate of the CYP3A4 pathway with a narrow therapeutic index

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12 week endpoint in glycosylated fraction of hemoglobin A (HbA1c) | Baseline, 12 Weeks

SECONDARY OUTCOMES:
Change from baseline to 12 week endpoint in fasting blood glucose | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in average Seven Point Self Monitored Blood Glucose | Baseline, 12 Weeks
Change from baseline to 12 week endpoint for Oral Glucose Tolerance Test (OGTT) | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in Homa-B: Insulin | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in Homa-IR: Insulin | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in Homa-S: Insulin | Baseline, 12 weeks
Change from baseline to 12 week endpoint in fasting lipids | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in free fatty acids | Baseline, 12 Weeks
Change from baseline to 12 week endpoint in body weight | Baseline, 12 Weeks
Incidence of Hypoglycemic Episodes | Baseline through 12 weeks
Percentage of participants at each dose level up to 12 weeks | Baseline up to 12 weeks
Pharmacokinetics: Maximum plasma concentration (Cmax) of LY2608204 | pre-dose, up to 12 hours post-dose
Number of participants with severe hypoglycemic episodes | Baseline through 12 weeks
Rate of hypoglycemic episodes | Baseline through 12 weeks
Pharmacokinetics: Area under the curve of concentration-time curve for one dosing interval at steady state (AUC0-tau, ss) of LY2608204 | pre-dose, up to 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perrysburg, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hurst, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plano, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vorarlberg
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Mergentheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Oeynhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giengen an der Brenz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petrel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville